CLINICAL TRIAL: NCT01101321
Title: A Randomized, Open-Label, Single-Dose, Two-Way Crossover Study in Healthy Subjects to Determine the Fasting Bioequivalence of Oxycodone Tamper Resistant (OTR) 80-mg Tablets Manufactured at the Totowa, NJ Facility to Oxycodone Tamper Resistant (OTR) 80-mg Tablets Manufactured at the Wilson, NC Facility
Brief Title: To Determine the Fasting Bioequivalence of Reformulated OXY Tablets Manufactured at Two Different Facilities
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Purdue Pharma LP (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: OTR1015
Record Dates: First submitted 2010-04-08; First posted 2010-04-09 (Estimated); Results first posted 2010-05-12 (Estimated); Last update posted 2015-11-18 (Estimated); Status verified 2015-10

CONDITIONS: Healthy
Keywords: Healthy subjects; Opioid; Healthy volunteers
MeSH Terms: interventions — Oxycodone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Reformulated OXY 80 mg (Totowa) (Experimental): Reformulated OXY 80 mg (Totowa) x 1 dose
  Interventions: Drug: Reformulated OXY (Totowa) (oxycodone HCl)
- Reformulated OXY 80 mg (Wilson) (Active Comparator): Reformulated OXY 80 mg (Wilson) x 1 dose
  Interventions: Drug: Reformulated OXY (Wilson) (oxycodone HCl)

INTERVENTIONS:
Drug: Reformulated OXY (Totowa) (oxycodone HCl) — Reformulated OXY 80-mg tablet (Totowa) x 1 dose taken without food.
  Arms: Reformulated OXY 80 mg (Totowa)
Drug: Reformulated OXY (Wilson) (oxycodone HCl) — Reformulated OXY 80-mg tablet (Wilson) x 1 dose taken without food.
  Arms: Reformulated OXY 80 mg (Wilson)

SUMMARY:
The purpose of this study is to assess the bioequivalence of a new oxycodone formulation (80 mg) manufactured at the Totowa, NJ facility relative to the formulation (80 mg) manufactured at the Wilson, NC facility in the fasted state.

DETAILED DESCRIPTION:
Oxycodone hydrochloride (oxycodone) is a semi-synthetic opioid analgesic that is effective in the relief of moderate to severe malignant and non-malignant pain.

ELIGIBILITY:
Inclusion Criteria:

* Males and females aged 18 to 50, inclusive.
* Body weight ranging from 50 to 100 kg and a BMI ≥18 and ≤34 (kg/m2).
* Healthy and free of significant abnormal findings as determined by medical history, physical examination, vital signs, and ECG.
* Females of child-bearing potential must be using an adequate and reliable method of contraception.

Exclusion Criteria:

* Females who are pregnant or lactating.
* Any history of or current drug or alcohol abuse for 5 years.
* History of or any current conditions that might interfere with drug absorption, distribution, metabolism or excretion.
* Use of an opioid-containing medication in the past 30 days.
* History of known sensitivity to oxycodone, naltrexone, or related compounds.
* Any history of frequent nausea or emesis regardless of etiology.
* Any history of seizures or head trauma with current sequelae.
* Participation in a clinical drug study during the 30 days preceding the initial dose in this study.
* Any significant illness during the 30 days preceding the initial dose in this study.
* Use of any medication including thyroid hormone replacement therapy (hormonal contraception is allowed), vitamins, herbal, and/or mineral supplements, during the 7 days preceding the initial dose.
* Refusal to abstain from food for 4 hours following administration of the study drugs and to abstain from caffeine or xanthine entirely during each confinement.
* Consumption of alcoholic beverages within forty-eight (48) hours of initial study drug administration (Day 1) or anytime following initial study drug administration.
* History of smoking or use of nicotine products within 45 days of study drug administration or a positive urine cotinine test.
* Blood or blood products donated within 30 days prior to administration of the study drugs or anytime during the study, except as required by this protocol.
* Positive results for urine drug screen or alcohol screen at Check-in of each period, and HBsAg, HBsAb (unless immunized), anti-HCV.
* Positive Naloxone HCl challenge test.
* Presence of Gilbert's Syndrome or any known hepatobiliary abnormalities.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 58 (Actual)
Dates: Start 2008-06; Primary Completion 2008-08 (Actual); Study Completion 2008-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Covance Clinical Research Unit Honolulu, Honolulu, Hawaii, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 23-Jun-2008 (first Informed Consent Form signed) to 19-Aug-2008 (last subject last visit), at 1 site in the US (Honolulu, HI).
Pre-assignment Details: 114 screened; 52 screen failures; 4 withdrew prior to randomization; 58 randomized; 8 terminated early; 50 completed.
Groups:
- Reformulated OXY (Totowa) (Test) First: Reformulated OXY 80-mg tablet (Totowa)(Test) fasted, dose administered in a two-period, two-sequence, single-dose, two-way crossover fashion. A minimum washout period of at least 6 days separated dose administrations. Subjects in this sequence received Reformulated OXY (Totowa) (Test) in period 1 and Reformulated OXY (Wilson) (Reference) in period 2.
- Reformulated OXY (Wilson) (Reference) First: Reformulated OXY 80-mg tablet (Wilson) (Reference) fasted, dose administered in a two-period, two-sequence, single-dose, two-way crossover fashion. A minimum washout period of at least 6 days separated dose administrations. Subjects in this sequence received Reformulated OXY (Wilson) (Reference) in period 1 and Reformulated OXY (Totowa) (Test) in period 2.
Period: Period 1
Arm/Group | Reformulated OXY (Totowa) (Test) First | Reformulated OXY (Wilson) (Reference) First
Started | 30 | 28
Completed | 26 | 24
Not Completed | 4 | 4
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Adverse Event | 3 | 3
Period: Period 2
Arm/Group | Reformulated OXY (Totowa) (Test) First | Reformulated OXY (Wilson) (Reference) First
Started | 26 | 24
Completed | 26 | 24
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Randomized Safety Population: Subjects who were randomized, received study drug, and had at least 1 postdose safety assessment.
Arm/Group | Randomized Safety Population
Number analyzed (Participants) | 58
Age, Continuous [Mean (Standard Deviation); unit: years] | 30 (9.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22
  Male | 36

OUTCOME MEASURES:

1. Primary Outcome: Cmax - Maximum Observed Plasma Concentration
Description: Bioequivalence based on Cmax
Time Frame: Blood samples collected over 72-hour period
Population: Full Analysis Population for PK Metrics. Data from all subjects who were randomized, received study drug, and had at least 1 valid PK metric variable were included in the statistical analysis.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Reformulated OXY (Totowa) (Test): Reformulated OXY 80-mg tablet (test) fasted, dose administered in a two-period, two-sequence, single-dose, two-way crossover fashion.
- Reformulated OXY (Wilson) (Reference): Reformulated OXY 80-mg tablet Wilson, NC (reference) fasted, dose administered in a two-period, two-sequence, single-dose, two-way crossover fashion.
Arm/Group | Reformulated OXY (Totowa) (Test) | Reformulated OXY (Wilson) (Reference)
Number analyzed (Participants) | 47 | 50
ng/mL | 78.4 (20.8) | 78.2 (20.2)
Statistical Analysis 1: Comparison: Reformulated OXY (Totowa) (Test) vs Reformulated OXY (Wilson) (Reference); Test type: Non-Inferiority or Equivalence — A mixed-model analysis of variance was used to compare (test vs reference) and the 90% confidence intervals were estimated for the ratios (test/reference); ANOVA; Geometric Test/Ref Ratio x 100 = 100, 90% CI 2-sided [96.14 to 104.96] — Bioequivalence is established when 90% Confidence Interval falls within 80%-125%

2. Primary Outcome: AUC0-inf - Area Under Plasma Concentration-time Curve From Time Zero to Infinity (Extrapolated)
Description: Bioequivalence based on AUC0-inf
Time Frame: Blood samples collected over 72-hour period
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Reformulated OXY (Totowa) (Test) | Reformulated OXY (Wilson) (Reference)
Number analyzed (Participants) | 47 | 50
ng*h/mL | 846 (223) | 850 (191)
Statistical Analysis 1: Comparison: Reformulated OXY (Totowa) (Test) vs Reformulated OXY (Wilson) (Reference); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; ANOVA; Geometric Test/Ref Ratio x 100 = 98.5, 90% CI 2-sided [95.44 to 101.73] — Bioequivalence is established when 90% Confidence Interval falls within 80%-125%

3. Primary Outcome: AUC0-t - Area Under Plasma Concentration-time Curve From Time Zero to Time of Last Non-zero Plasma Concentration
Description: Bioequivalence based on AUC0-t
Time Frame: Blood samples collected over 72-hour period
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Reformulated OXY (Totowa) (Test) | Reformulated OXY (Wilson) (Reference)
Number analyzed (Participants) | 47 | 50
ng*h/mL | 843 (223) | 848 (191)
Statistical Analysis 1: Comparison: Reformulated OXY (Totowa) (Test) vs Reformulated OXY (Wilson) (Reference); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; ANOVA; Geometric Test/Ref Ratio x 100 = 98.5, 90% CI 2-sided [95.42 to 101.70] — Bioequivalence is established when 90% Confidence Interval falls within 80%-125%

ADVERSE EVENTS:
Time Frame: Ongoing AEs-followed until resolution/30 days after last dose;AEs reported during 7 days following last dose were recorded & followed until resolution or up to 30 days after last dose. All SAEs were followed until resolution or event/sequelae stabilized.
Description: AEs were learned of through spontaneous reports, subject interview, or subject diaries.
Arm/Group | Reformulated OXY (Totowa) (Test) | Reformulated OXY (Wilson) (Reference)
Serious Adverse Events (participants affected / at risk) | 0/54 | 0/54
Other Adverse Events (participants affected / at risk) | 29/54 | 22/54
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Reformulated OXY (Totowa) (Test) (N=54) | Reformulated OXY (Wilson) (Reference) (N=54)
Abdominal Pain (Gastrointestinal disorders) | 4 (4) | 6 (6) — Systematic and nonsystematic assessments were used for reporting AEs.
Nausea (Gastrointestinal disorders) | 11 (16) | 7 (7) — Systematic and nonsystematic assessments were used for reporting AEs.
Vomiting (Gastrointestinal disorders) | 8 (18) | 8 (19) — Systematic and nonsystematic assessments were used for reporting AEs.
Fatigue (General disorders) | 3 (3) | 4 (4) — Systematic and nonsystematic assessments were used for reporting AEs.
Dizziness (Nervous system disorders) | 8 (10) | 6 (8) — Systematic and nonsystematic assessments were used for reporting AEs.
Headache (Nervous system disorders) | 13 (14) | 8 (11) — Systematic and nonsystematic assessments were used for reporting AEs.
Somnolence (Nervous system disorders) | 11 (12) | 5 (5) — Systematic and nonsystematic assessments were used for reporting AEs.
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 4 (4) — Systematic and nonsystematic assessments were used for reporting AEs.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days